CLINICAL TRIAL: NCT03212443
Title: Combined Suprascapular and Axillary Nerve Blocks for Sevoflurane Consumption and Postoperative Analgesia in Arthroscopic Shoulder Surgery
Brief Title: Combined Suprascapular and Axillary Nerve Blocks for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Associated professor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diskapi4
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Arthroscopic Shoulder Surgery; Suprascapular Nerve Block; Axillary Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Sham Comparator): In group A, the surgeon will apply 20 ml of 0.250% bupivacaine to the subacromial region at the end of the procedure
  Interventions: Procedure: Subacromial infiltration
- Group B (Active Comparator): In Group B, suprascapular (10 ml of 0.250% bupivacaine ) and axillary block (10 ml of 0.250% bupivacaine) will be performed with ultrasound and nerve stimulator guidance before induction of anesthesia
  Interventions: Procedure: Suprascapular nerve- axillary nerve block combination

INTERVENTIONS:
Procedure: Suprascapular nerve- axillary nerve block combination — In Group B, suprascapular (10 ml of 0.250% bupivacaine ) and axillary block (10 ml of 0.250% bupivacaine) will be performed with ultrasound and nerve stimulator guidance before induction of anesthesia
  Arms: Group B
Procedure: Subacromial infiltration — In group A, the surgeon will apply 20 ml of 0.250% bupivacaine to the subacromial region at the end of the procedure
  Arms: Group A

SUMMARY:
Arthroscopic shoulder surgery is associated with severe pain postoperatively. Regional nerve block adding to general anesthesia might improve the quality of postoperative analgesia. The aim of the study is to compare the subacromial local anesthetic infiltration and the suprascapular-axillary nerve blocks combination for intraoperative sevoflurane consumption, postoperative analgesia and analgesic consumption.

DETAILED DESCRIPTION:
After informed consent and with ethics approval, 60 ASA 2-3 patients scheduled for elective arthroscopic shoulder surgery will be included in this study. Patient will be divided to two groups by using computer -generated list for randomization. In group A, the surgeon will apply 20 ml of 0.250% bupivacaine to the subacromial region at the end of the procedure. In Group B, suprascapular (10 ml of 0.250% bupivacaine ) and axillary block (10 ml of 0.250% bupivacaine) will be performed with ultrasound and nerve stimulator guidance before induction of anesthesia. In all patients after standard and BIS (Bi spectral index) monitorization general anesthesia will be induced with remifentanil (10mcg iv), propofol (2.5 mg/kg iv) and rocuronium (0.5mg/kg iv). After intubation, anesthesia will be maintained with 50% O2 and N2O mixture. Hemodynamic parameters, BIS values, end-tidal sevoflurane consumption will be recorded by blind investigator. Postoperative visual analog scale (VAS) values, postoperative analgesic consumption (Tramadol, patient controlled analgesia), complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesia physical status (ASA) 1,2 patients
* Elective arthroscopic shoulder surgery

Exclusion Criteria:

* ASA 3,4 patients
* Coagulation abnormality
* Body mass index >30
* Preexisting neurological deficit Local anesthetic allergy history Diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Postoperative VAS scores | Through postoperative period, an avarage of 30 minutes
  Ranging from 0: no pain to 10: worst pain

SECONDARY OUTCOMES:
sevoflurane consumption | 5th, 10th,20th,30th,40th,50th minutes after induction of anesthesia
  End tidal sevoflurane concentration values assesment during the surgery

OTHER OUTCOMES:
Bleeding assesment | 5th, 10th,20th,30th,40th,50th minutes after induction of anesthesia
  stage1: Good surgical visualization (numeric rating scale 7<), Stage 2: Moderate bleeding (numeric rating sacle =4-7), Stage 3: Severe bleeding, bad surgical visualization (numeric rating scale < 4)

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozkan, Principal Investigator — Ministry of Health Diskapi Yildirim Beyazit Training and Research Hospital
Locations (1):
- Derya Ozkan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhir S, Sondekoppam RV, Sharma R, Ganapathy S, Athwal GS. A Comparison of Combined Suprascapular and Axillary Nerve Blocks to Interscalene Nerve Block for Analgesia in Arthroscopic Shoulder Surgery: An Equivalence Study. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):564-71. doi: 10.1097/AAP.0000000000000436. PMID 27380105
- [Result] Ritchie ED, Tong D, Chung F, Norris AM, Miniaci A, Vairavanathan SD. Suprascapular nerve block for postoperative pain relief in arthroscopic shoulder surgery: a new modality? Anesth Analg. 1997 Jun;84(6):1306-12. doi: 10.1097/00000539-199706000-00024. PMID 9174311